CLINICAL TRIAL: NCT01528722
Title: Double Blind Sham Controlled Randomised Trial of Intraperitoneal Bupivacaine During Acute Laparoscopic Cholecystectomy
Brief Title: Randomized Control Trial of Intraperitoneal Bupivacaine During Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Keith Roberts, Mr, University Hospitals Coventry and Warwickshire NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Acute lap chole RCT
Record Dates: First submitted 2012-02-04; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Cholecystitis; Gall Stone Pancreatitis
Keywords: Emergency laparoscopic cholecystectomy; Pain scores; Intraperitoneal local anaesthesia; Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline sham injection (Sham Comparator): Sham wash and injection with normal saline (09%)
  Interventions: Other: Normal saline
- Bupivacaine (Active Comparator): Bupivacaine injection/wash treatment arm
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.25% 20ml administered intraperitoneal
  Other Names: Marcaine
  Arms: Bupivacaine
Other: Normal saline — sodium chloride 0.9% solution
  Arms: Saline sham injection

SUMMARY:
Laparoscopic cholecystectomy (removal of the gall bladder via 'keyhole surgery') is a common procedure. This can be performed as an emergency operation when a patient has a complication of gall stones such as acute inflammation or pancreatitis. There are several trials which demonstrate that placing local anaesthetic inside the abdomen at the site of gall bladder surgery during a planned elective operation decreases post operative pain. This is the first trial to investigate the efficacy of this local anaesthetic during emergency cholecystectomy.

DETAILED DESCRIPTION:
Background Several studies, including a metanalysis, have demonstrated that intraperitoneal local anaesthetic (IP LA) during elective laparoscopic cholecystectomy (el-LC) decreases post operative pain. None have explored the efficacy of IP LA at emergency laparoscopic cholecystectomy (em-LC). A longer operation duration, greater frequency of washing and the inflammation associated with cholecystitis or pancreatitis are a few reasons why it cannot be assumed that a benefit in pain scores will be seen in em-LC with IP LA. This study assesses the efficacy of IP LA used in patients undergoing em-LC.

Methods Double blind randomised sham controlled trial of 42 consecutive subjects undergoing em- LC.

IP-LA was delivered by a combination of direct injection to the diaphragmatic and topical wash over the liver/gall bladder with bupivacaine or sham depending upon allocation. The primary outcome was VAS pain scores on the ward. Secondary outcomes included VRS pain scores in theatre recovery, analgesic use, physiological observations, time to eating and ambulation and length of postoperative stay.

Results One patient had a procedure converted to open and was excluded. There was no significant difference in pain scores on the ward or in theatre recovery. Analgesic use, respiratory rate, oxygen saturation, duration to ambulation, eating, satisfaction scores and time to discharge were comparable between the groups.

Conclusions Intraperitoneal LA during em-LC does not influence post-operative pain. Other modalities of analgesia should be explored as well as decreasing the interval between diagnosis of acute admission and em-LC.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing emergency cholecystectomy for cholecystitis or gall stone pancreatitis

Exclusion Criteria:

* patients undergoing planned elective cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
VAS pain score

SECONDARY OUTCOMES:
VRS pain score
Satisfaction score (VAS)
Physiological observations - respiratory rate, oxygen saturation
Analgesic use post operation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry and Warwickshire, Coventry, Warwickshire, United Kingdom

REFERENCES:
- [Derived] Roberts KJ, Gilmour J, Pande R, Hodson J, Lam FT, Khan S. Double-blind randomized sham controlled trial of intraperitoneal bupivacaine during emergency laparoscopic cholecystectomy. Hepatobiliary Pancreat Dis Int. 2013 Jun;12(3):310-6. doi: 10.1016/s1499-3872(13)60049-1. PMID 23742777